CLINICAL TRIAL: NCT00282893
Title: Balloon Prophylaxis of Aneurysmal Vasospasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 200311385; R01NS038484 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2014-03

CONDITIONS: Aneurysm; Vasospasm
Keywords: aneurysm; vasospasm; subarachnoid hemorrhage; transluminal ballooning
MeSH Terms: conditions — Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pTBA (Experimental): Prophylactic Transluminal Ballooning Angioplasty
  Interventions: Procedure: transluminal ballooning
- Control (Active Comparator): currently existing therapies for the treatment of vasospasm
  Interventions: Other: currently existing therapies for the treatment of vasospasm

INTERVENTIONS:
Procedure: transluminal ballooning
  Arms: pTBA
Other: currently existing therapies for the treatment of vasospasm
  Arms: Control

SUMMARY:
The purpose of this study is to determine if early transluminal ballooning of the major cerebral arteries prevents severe vasospasm and improves neurological outcome in patients with Fisher Grade III aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (SAH) afflicts over 30,000 patients a year in the United States. Fifteen percent of those who survive the initial bleeding die or suffer disabilities because of delayed ischemic deficit (stroke) due to vasospasm. Vasospasm is a condition in which the arteries in the brain constrict, not allowing sufficient blood flow and oxygenation. Research on the pharmacological prevention and treatment of vasospasm has resulted in only minimal improvement for this problem.

Transluminal ballooning is a procedure that opens blood vessels, allowing blood flow and oxygen to get to the brain more easily. Researchers believe that this dilation of the blood vessels lasts for at least 7 days. This procedure is used to treat severe vasospasm although it is not commonly used to prevent vasospasm. The purpose of this trial is to find out if this procedure, performed immediately after the aneurysm is secured, prevents spasm in the brain and improves patient outcome.

Eligible SAH patients whose aneurysm has been repaired by neurosurgical or endovascular procedure and who are enrolled in the study will be randomized to receive either the prophylactic transluminal ballooning procedure or to receive standard care, which includes currently existing therapies for the treatment of vasospasm.

Participants will be asked to return for follow-up examinations at 3 and 6 months to evaluate recovery using a standardized outcome scale.

ELIGIBILITY:
Inclusion Criteria:

* Fisher grade III hemorrhage
* Documented ruptured cerebral aneurysm via angiography, CT angiogram or any other acceptable neuroradiologic means
* Ruptured aneurysm(s) secured
* Ballooning available < 96 hours post SAH

Exclusion Criteria:

* Vasospasm prior to randomization
* Interventionalist unavailable
* Patient outside the 96 hour window for ballooning
* Enrolled in competing trial
* Unsecured aneurysms (symptomatic or asymptomatic) that are in the location where the ballooning procedure would occur
* Medical conditions known that would effect mortality / morbidity
* Severe Cerebrovascular atherosclerosis
* > 16 years old.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2000-10; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Dichotomized Glasgow Outcome Scale (GOS)assessed at 3 months by a blinded evaluator

SECONDARY OUTCOMES:
Dichotomized GOS at 6 months, assessment at 3 and 6 months of: five-point GOS; GOS - Extended (GOSE), occurrence of delayed ischemic deficit (DID), the incidence of severe vasospasm as detected by Transcranial Doppler (TCD) Ultrasonography (mean blood f

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Muizelaar, MD, PhD, Principal Investigator — Professor and Chairman, Department of Neurological Surgery, University of California, Davis; Jonathan Hartman, MD, Principal Investigator — Interventional Neuroradiologist, University of California, Davis; Marike Zwienenberg, MD, Principal Investigator — University of California, Davis
Locations (5):
- United States (3):
  - Coordinating Center: University of California, Davis Medical Center, Department of Neurological Surgery, Sacramento, California
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington - Harborview Medical Center, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada
- University Medical Center Utrecht, Trialbeureau Neurodivisie, Heidelberglaan 100, Utrecht, Netherlands

REFERENCES:
- [Result] Zwienenberg-Lee M, Hartman J, Rudisill N, Madden LK, Smith K, Eskridge J, Newell D, Verweij B, Bullock MR, Baker A, Coplin W, Mericle R, Dai J, Rocke D, Muizelaar JP; Balloon Prophylaxis for Aneurysmal Vasospasm (BPAV) Study Group. Effect of prophylactic transluminal balloon angioplasty on cerebral vasospasm and outcome in patients with Fisher grade III subarachnoid hemorrhage: results of a phase II multicenter, randomized, clinical trial. Stroke. 2008 Jun;39(6):1759-65. doi: 10.1161/STROKEAHA.107.502666. Epub 2008 Apr 17. PMID 18420953